CLINICAL TRIAL: NCT03154021
Title: Clinical Effectiveness of Next Science Oral Rinse in Controlling Plaques and Gingival Inflammation
Brief Title: Next Science Antimicrobial Mouth Rinse Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Next Science LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB201700505; CSP-007 (Other: University of Florida)
Record Dates: First submitted 2017-05-05; First posted 2017-05-15 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Gingivitis; Dental Plaque
Keywords: Gingival Index; Plaque Index; Bleeding; Pocket Depth
MeSH Terms: conditions — Gingivitis; Dental Plaque; Hemorrhage | interventions — Oils, Volatile

STUDY DESIGN:
Intervention Model Description: One half of subjects will be given test product other half will be given placebo.
Who Masked: Participant, Investigator
Masking Description: The identity of the experimental oral rinse and its placebo will be disguised. Test and control kit boxes will contain toothpaste, a toothbrush, dose cups and a timer. The kit boxes will be labeled with a unique kit number representing the test product or placebo known only to the manufacturer. Kit box labels will also contain the study number, emergency phone number, distributor name/address, appropriate caution statements, content statement and other information as required by internal regulations and clinical SOPs. Kit box content statement will be worded to maintain the study blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gingivitis Test (Experimental): All subjects will have oral examination, dental cleaning, plaque samples taken, given Colgate Total Toothpaste, Oral B Manual Toothbrush and Next Science Over the Counter (OTC) Oral Rinse with Essential Oils.
  Interventions: Combination Product: Next Science OTC Oral Rinse with Essential Oils
- Gingivitis Placebo (Placebo Comparator): All subjects will have oral examination, dental cleaning, plaque samples taken, given Colgate Total Toothpaste, Oral B Manual Toothbrush and OTC Oral Rinse Control.
  Interventions: Combination Product: OTC Oral Rinse Control

INTERVENTIONS:
Combination Product: Next Science OTC Oral Rinse with Essential Oils — This group will receive Next Science Oral Rinse with Essential Oils and the other half will be give OTC Oral Rinse Control
  Arms: Gingivitis Test
Combination Product: OTC Oral Rinse Control — This group will receive OTC Oral Rinse Control
  Arms: Gingivitis Placebo

SUMMARY:
To assess the effect of a test antimicrobial oral rinse from Next Science on the prevention of oral biofilm formation and thereby preventing gingivitis by monitoring the oral microbial flora and measuring gingival inflammation and bleeding.

DETAILED DESCRIPTION:
Baseline, Visit 1:

Prior to this visit subjects will be asked not to perform any oral hygiene the morning of the visit. They will also be asked not to use medicated lozenges, breath mints, toothpicks, eat, drink (except water), smoke and/or chew gum the morning of the study visit. Subjects will be asked to read and sign an informed consent and they will be given a signed copy. Personal medical history information will be reviewed and retained as site source documentation. Demographic Information and entrance criteria will be assessed. A comprehensive oral examination will then be conducted to evaluate the oral and perioral region, including hard and soft tissues. This will include periodontal charting for pocket depths, plaque scores as well as gingival index and bleeding scores. Plaque samples will be collected from the following four sites- mesial surface of maxillary first molar on left side, distal surface of maxillary first premolar on right side, mesial surface of mandibular second molar on left side and distal surface of mandibular lateral incisor on right side. If any of these four teeth are missing, the next tooth mesial to it will be used to collect the plaque sample.

Visit 2: Dental Prophylaxis, Oral Hygiene Instruction and Product Dispensation Subjects will receive a whole-mouth dental prophylaxis by the dental hygienist. For logistical reasons, the Dental Prophylaxis visit may occur within 2 weeks of the Baseline Visit. This visit will also include instructions on oral hygiene, dispensation of tooth brush/toothpaste and the oral rinse product. The experimental oral rinse product and the placebo will be provided by the manufacturer fully coded in prepacked bottles with the code numbers. Subjects will be instructed to brush their teeth and rinse their mouth with the dispensed product twice daily (AM/PM) for 30 seconds. A sheet of paper with pre-marked dates will be provided to each subject for them to record the time of the day they rinsed and duration. Subjects will be asked not to perform any oral hygiene the morning of their next visit. They will also be asked not to use medicated lozenges, breath mints, toothpicks, eat, drink (except water), smoke and/or chew gum the morning of the next study visit.

Week 6, Visit 3:

Subjects will be asked if they have performed any oral hygiene the morning of the visit. They will also be asked if they have used medicated lozenges, breath mints, toothpicks, eaten, had anything to drink (other than water), smoked and/or chewed gum the morning of the study visit. The paper sheet with recording of their rinsing habits will be collected. An oral examination will be conducted, an assessment of plaques and gingival scores will occur with periodontal charting for pocket depths, plaque scores as well as gingival index and bleeding scores. Dental plaque samples will be collected as before from the same sites. Any untoward experiences and findings will be recorded (example- change in taste sensation, any ulcers, blisters, etc.). New paper sheet to document their daily use of oral rinse will be provided. Subjects will be asked not to perform any oral hygiene the morning of their next visit. They will also be asked not to use medicated lozenges, breath mints, toothpicks, eat, drink (except water), smoke and/or chew gum the morning of the next study visit.

Week 12, Visit 4:

Subjects will be asked if they have performed any oral hygiene the morning of the visit. They will also be asked if they have used medicated lozenges, breath mints, toothpicks, eaten, had anything to drink (other than water), smoked and/or chewed gum the morning of the study visit.

The paper sheet with recording of their rinsing habits will be collected. Full mouth periodontal charting to include plaque and bleeding scores as well as gingival index will be recorded and dental plaque samples collected as before (from the same sites). Any untoward experiences and findings will be recorded (example- change in taste sensation, any ulcers, blisters, etc.). Patients will be informed of any dental treatment needs and general comments and Adverse Events, if applicable, will be recorded. A subject accountability form will be completed and subjects will be dismissed from the study. A subject accountability form will also be completed for subjects who drop out of the study prior to its completion.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 60
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form (ICF).
* Be in good general health as determined by the investigator/designee based on a review of the Medical history/update for participation in the study;
* Have at least 20 gradable teeth;
* Have 10 or more bleeding sites at Baseline

Exclusion Criteria:

* Known allergies or sensitivity to oral rinse products, especially those containing cetylpyridinium chloride (CPC), sodium hydroxide or potassium dihydrogen phosphate.
* Severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession.
* Active treatment for periodontitis.
* Braces
* Diabetes
* Antibiotic use within three months of the Baseline, Visit 1.
* Pregnancy
* Any diseases or conditions that could be expected to interfere with the subject safely completing the study.

Continuance Criteria

Subjects may be excluded from the study or the analysis due to:

* Use of antibiotics any time during the study;
* Use of any non-study oral hygiene products during the study;
* A non-study dental prophylaxis or other elective dentistry during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-03-08 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Oral Exam to see if there are any changes in pocket depths at two weeks, six weeks and twelve weeks | Baseline, six weeks and twelve weeks.
  Complete oral exam with charting of pocket depths
Gingival Index to see if there are any changes in gingival index at two weeks, six weeks and twelve weeks. | Baseline, six weeks and twelve weeks.
  Gingival Index using Loe and Silness Gingival index
Plaque index to see if there are any changes in plaque scores at two weeks, six weeks and twelve weeks. | Baseline, six weeks and twelve weeks
  Plaque index using Turesky Plaque Index
Bleeding Scores to see if there are any changes in bleeding at two weeks, six weeks and twelve weeks. | Baseline, six weeks and twelve weeks.
  Check for bleeding sites

SECONDARY OUTCOMES:
Plaque samples to see if there is any change in samples at two weeks, six weeks, and twelve weeks. | Baseline, six weeks and twelve weeks.
  Plaque samples will be collected from the following four sites- mesial surface of maxillary first molar on left side, distal surface of maxillary first premolar on right side, mesial surface of mandibular second molar on left side and distal surface of mandibular lateral incisor on right side. These samples will be analyzed for composition of oral microbial flora.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Progulske-Fox, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Dental Clinical Research Unit, University of Florida, Gainesville, Florida
  - University of Florida College of Dentistry, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Newman BA, Rosebrough CN, Tamashiro RA, Dias Ribeiro AP, Whitlock JA, Sidhu G, Aukhil I, Porral DY, Progulske-Fox A, Myntti MF, Wang GP. A randomized controlled trial to evaluate the effectiveness of a novel mouth rinse in patients with gingivitis. BMC Oral Health. 2022 Nov 2;22(1):461. doi: 10.1186/s12903-022-02518-2. PMID 36324127